CLINICAL TRIAL: NCT00650403
Title: Single-Dose Fed Bioequivalence Study of Paroxetine Hydrochloride Tablets (40 mg; Mylan) and Paxil® Tablets (40 mg; GSK) in Healthy Adult Volunteers
Brief Title: Food Study of Paroxetine Hydrochloride Tablets 40 mg and Paxil® Tablets 40 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PARO-0679
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Paroxetine; Tablets

ARMS (2):
- 1 (Experimental): Paroxetine hydrochloride 40 mg tablet
  Interventions: Drug: Paroxetine hydrochloride 40 mg tablet
- 2 (Active Comparator): Paxil® 40 mg Tablet
  Interventions: Drug: Paxil® 40 mg Tablet

INTERVENTIONS:
Drug: Paroxetine hydrochloride 40 mg tablet — 40mg, single dose fed
  Arms: 1
Drug: Paxil® 40 mg Tablet — 40mg, single dose fed
  Arms: 2

SUMMARY:
The objective of this study is to investigate the bioequivalence of Mylan's paroxetine hydrochloride 40 mg tablets to GSK's Paxil® 40 mg tablets following a single, oral 40 mg (1 x 40 mg) dose administered under fed conditions to healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who were informed of the nature of the study and agreed to read, review, and sign the informed consent document prior to Period I dosing.
2. Subjects who completed the screening process within 21 days prior to Period I dosing.
3. Subjects who were healthy adult men and women at least 18 years of age at the time of dosing.
4. Subjects who weighed at least 60 kg (132 lbs) for men and 48 kg (106 lbs) for women. All subjects must have a Body Mass Index (BMI) less than or equal to 30 but greater than or equal to 19.
5. Subjects who were healthy as documented by the medical history, physical examination (including but not limited to an evaluation of the cardiovascular, gastrointestinal, respiratory, and central nervous systems), vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and by general observations. Any abnormalities/deviations from the normal range which was considered clinically relevant by the study physician and investigator was evaluated for individual cases, documented in study files, and agreed upon by the investigator and clinic personnel prior to enrolling a volunteer in this study and for continued enrollment.
6. Subjects who had a negative urine drug screen.
7. Female subjects who had a negative pregnancy screen.
8. Female subjects were physically incapable of pregnancy - surgically sterile (bilateral oophorectomy with an absence of bleeding for six months, with or without a hysterectomy, or total hysterectomy and an absence of bleeding for at least three months) or post-menopausal with an absence of menses for at least 12 months.
9. During the course of the study, from study screen until study exit - including the washout period, all men used a spermicide containing barrier method of contraception.

Exclusion Criteria:

1. Institutionalized subjects were not used.
2. Social Habits: a. Use of any tobacco-containing products within one (1) year prior to dosing. b. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication. c. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication. d. Any recent, significant change in dietary or exercise habits. e. A positive test for any drug included in the urine drug screen. f. History of drug and/or alcohol abuse.
3. Medications: a. Use of any prescription or over-the-counter (OTC) medication within the 14 days prior to the initial dose of study medication. b. Use of any hormonal contraceptives or hormone replacement therapy within 3 months prior to study medication dosing. c. Use of any medication within 28 days prior to initial dose of study medication unless the Pharmacokinetics/Drug Metabolism Department at Mylan was consulted and a decision was made to allow the subjects to enroll based on the medications pharmacology and pharmacokinetics. d. Use of monoamine oxidase inhibitors (MAOIs), pimozide, or thioridazine within 30 days prior to the initial dosing of study medication.
4. Diseases: a. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, or neurologic disease. b. Acute illness at the time of either the pre-study medical evaluation or dosing. c. A positive HIV, hepatitis B, or hepatitis C test.
5. Abnormal and clinically significant laboratory test results: a. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities. b. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to paroxetine or other related products.
9. History of difficulties swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within seven (7) days of drug administration.
11. History of depression, mania, seizure, akathisia, narrow angle glaucoma, and/or suicidal ideation or behavior (suicidality).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruce T Czarnik, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html